CLINICAL TRIAL: NCT06843603
Title: Barriers/Facilitators and Care Coordination of Native Hawaiians & Kidney Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: National Kidney Foundation, United States (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 40709
Record Dates: First submitted 2025-02-13; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Kidney Disease, Chronic
Keywords: kidney disease, chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: We propose a mixed method design study with the goal to improve CKD rescreening among early stage high-risk NHs by aligning health equity with a culturally informed care coordination systems model. Guided by the CFIR 2.017, in Aim 1/Year 1 we will conduct a formative evaluation on the barriers and facilitators associated with increasing individual patient follow-up with their PCP after the initial NKFH KEDS screening and develop implementation strategies. Then in Aim 2/Year 2 we will examine the acceptability and feasibility of a selected culturally-informed care coordination intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Culturally Informed Care Coordination (Experimental): In this ARM, we will trial the culturally informed care coordination intervention to see if improves patient care follow-up
  Interventions: Behavioral: culturally informed care coordination intervention; Other: No Intervention - Usual Care Group
- Usual Care Group (No Intervention): In this Arm the Usual Care Group does not have an intervention.

INTERVENTIONS:
Behavioral: culturally informed care coordination intervention — Culturally Informed Care Coordination Strategies
  Arms: Culturally Informed Care Coordination
Other: No Intervention - Usual Care Group — No Intervention - Usual Care Group
  Arms: Culturally Informed Care Coordination

SUMMARY:
Native Hawaiians (NH) are 9.5 times more likely to be on dialysis or need a kidney transplant compared to Whites. They have the highest end-stage kidney disease (ESKD) incidence rates in the nation, begin dialysis at younger ages (30-50 years), and one of the most under-studied racial/ethnic groups in chronic kidney disease (CKD) research. This project's outcome is to improve kidney disease follow-up among early stage NHs at high risk by aligning health equity with a culturally appropriate care coordination systems model.

DETAILED DESCRIPTION:
SPECIFIC AIMS Native Hawaiians (NH) are 9.5 times more likely to be on dialysis or need a kidney transplant as compared to those who identify race as White. NH have the highest rates of end-stage kidney disease in the United States (US) and begin dialysis at younger ages (30-50 years). NHs are also at high risk for diabetes, hypertension, cardiovascular disease, stroke, & obesity which intersects with kidney disease. NHs are also one of the most under-studied racial/ethnic groups in chronic kidney disease (CKD) research.4 Therefore, there is a is critical need to examine and address kidney health disparities and inequities in the NH population.

This multi-disciplinary scientific team has conducted cross-sectional epidemiological early CKD studies over a 10-year period of time among NHs who participated in the National Kidney Foundation of Hawaii (NKFH) Kidney Early Detection & Screening (KEDS) Program. Our findings indicate NHs have a heightened risk of end stage kidney disease based on biological and clinical risk factors5 using CKD biomarkers (i.e. lab tests for estimated glomerular filtration rate (eGFR↓) and urinary albumin creatinine ratio (UACR↑). These tests are indicators of abnormal kidney function and damage. One of the US Healthy People 2030 goals is to increase the proportion of older adults with CKD to obtain recommended screening tests (eGFR, UACR) to identify CKD in the early stages. The NKFH KEDS program provides a comprehensive community early detection screening program where participants are sent their screening lab results and are asked to share these results with their primary care provider (PCP). Our previous research has highlighted significant gaps related to participant follow-up with their PCP. Therefore, using the NIMHD Framework adapted to reflect social and cultural influences of NH health focused on family and community support/resources, access to cultural institutions and practice, and access to services to optimal health and well-being, the overall goal of this study is to develop a culturally-informed care coordination model between NKFH KEDS NH participants and NKFH and PCP staff to improve screening follow-up. Our central hypothesis is that a theoretically-driven, culturally-informed, care coordination model will not improve follow-up for eGFR & UACR. To address this gap, this innovative study aims to adapt the abridged version of the Consolidated Framework for Implementation Research 2.0 framework named pragmatic context assessment tool (pCAT) for screening (eGFR, UACR) follow-up among NH adults in early stages of CKD. Specific Aims include:

Aim 1: Understand barriers and facilitators associated with culturally informed care coordination and follow-up for eGFR & UACR. First, we will conduct a formative evaluation on the barriers & facilitators of NKFH KEDS NH participants (n=25) and NKFH (n=15) and PCP (n=10) staff) and reach consensus by all (NH participants, NKFH and PCP staff, and a NH advisory group) of a feasible intervention - (1) NKFH KEDS NH participants, using the pCAT survey and interview and (2) NKFH and PCP staff, using the same pCAT18 survey and interview. NH participants (n=25) will be: (1) aged 18 years and older, (2) with eGFR < 60 ml/min/1.73m2 (Stage 3a-3b CKD) and/or ≥30 UACR, (3) have participated in the NKFH KEDS Program within 3 months, and (4) able to read, write, and speak English. NKFH (n=15) and PCP (n=10) staff's inclusion criteria include: (1) able to read, write & speak English and (2) aged 18 years and older. Three PCP sites will be selected due to high enrollment of NH patients in their practice. Consensus of key barriers/facilitators and contextual factors that will drive the intervention selection will be completed based on the evaluation results. The research team will summarize the literature on the implementation strategies, suggest strategies and reach consensus for a selected intervention by the end of study year 1. The advisory group will be made up of members from 3 NH non-profit organizations. Quantitative and qualitative analysis for the evaluation will be completed.

Aim 2: Examine the acceptability and feasibility of a culturally-informed care coordination intervention. Second, we will evaluate our intervention by selecting one PCP site to receive usual care and other PCP site will receive the culturally informed care coordination intervention. The NKFH KEDS NH participants (n=25) and NKFH (n=5) and PCP (n=5) staff (for each, control and intervention group) will be interviewed using the pCAT18 individual survey and interview evaluation and outcomes20 of our intervention in the first 6 months of study year 2. Finally, both quantitative and qualitative analysis will be used to examine the acceptability and feasibility of the intervention in the second half of year 2.

The long-term goal of this project is to improve CKD rescreening among early stage high-risk NHs by aligning health equity with a culturally appropriate care coordination systems model. To reach this goal, results from this NIH R21 project will provide the foundation for a pilot study for an NIH R34 IRINAH. This project has the potential for dissemination to other primary care provider offices and organizations - federally qualified community centers, and hospital clinics to increase re-screening rates among high risk NHs in the early stages of CKD between community and primary care provider follow-up.

ELIGIBILITY:
AIM 1 and AIM 2: Inclusion Criteria: Native Hawaiian (NH) participants from the NKFH KEDS program are:

* greater or equal to 18 years
* self-reported as Native Hawaiian
* eGFR less than 60 ml/min/1.73m2 (Stage 3a-3b CKD) and/or greater or equal to 30 mg/g UACR
* have participated in the NKFH KEDS Program within 3 months
* able to read, write, and speak English.

AIM 1 and AIM 2: Inclusion Criteria: NKFH and PCP staff are :

* able to read, write, and speak English,
* greater or equal to 18 years.

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability to Intervention | 9 months
  Acceptability (the degree to which an intervention is perceived a good fit)
  Acceptability will be measured by a survey likert scale of 1 (not acceptable) - 10 (most acceptable)
  Name of measurement tool is reference in Procter et al (p. 69):
  Procter E, Silmere H, Raghavan R, et al. Outcomes for implementation research, conceptual distinctions, measurement challenges, and research agenda. Adm Policy Mental Health. 2022: 38 (2): 65-76.
Adoption of the Intervention | 9 months
  Adoption (intent to implement)
  Adoption will be scored as 0 (not at all implemented), 5 (somewhat implemented), and 10 (fully implemented).
  Name of measurement tool is reference in Procter et al (p. 69):
  Procter E, Silmere H, Raghavan R, et al. Outcomes for implementation research, conceptual distinctions, measurement challenges, and research agenda. Adm Policy Mental Health. 2022: 38 (2): 65-76.
Feasibility of the Intervention | 9 months
  Feasibility (possibility of successful implementation),
  Feasibility will be measured by a survey likert scale of 1 (not feasible) - 10 (most feasible).
  Name of measurement tool is reference in Procter et al (p. 69):
  Procter E, Silmere H, Raghavan R, et al. Outcomes for implementation research, conceptual distinctions, measurement challenges, and research agenda. Adm Policy Mental Health. 2022: 38 (2): 65-76.

SECONDARY OUTCOMES:
Beliefs to Change of the Intervention | 9 months
  TOTAL SCORE of 4 Questions will measure the secondary outcome measure - Beliefs to Change.
  Believe that rescreening for eGFR & UACR can directly influence your health Believe that integrating eGFR and UACR are worthwhile use of health care services Believe that primary care providers are committed to supporting rescreening for eGFR & UACR Believe that rescreening for eGFR and UACR belong in primary care health services.
  Asked to complete a survey with a 10-point Likert scale (0=Strongly Disagree to 10=Strongly Agree). Scores will be added to obtain a Total Score to measure the secondary outcome measure - Beliefs to Change.

CONTACTS AND LOCATIONS:
Overall Officials: Merle R Kataoka-Yahiro, DrPH., MPH., MS., Principal Investigator — University of Hawaii at Manoa
Locations (1):
- National Kidney Foundation of Hawaii, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: Yes
A database will be established to store project data. Presentations, abstracts, and manuscripts related to the work will also be centrally stored. Once the project is finished and all analyses are complete, it is our intention to make public the clean study data set (while maintaining the integrity of intellectual property and ensuring confidentiality of all human subjects clinical data). This data will be free of identifiers that will permit linkages to individual research participants and variable that could lead to disclosure of the identity of individual subjects. Investigators wishing to use the data will submit a written request to the contact PI and provide a data use agreement with University of Hawaii at Manoa and National Kidney Foundation of Hawaii. We will make the data and associated documentation available to users only under a data-sharing agreement with terms has been approved and signed.
Supporting Information: Study Protocol, SAP
Time Frame: New data from AIM 1 and 2 will be to NIH no later than 12 months after the award begins or at the time of publication of the first manuscript from this study. Scientific data included in published manuscripts will be make available at the time of publication, all other data will be made available no later than the end of the award. Data will be preserved and available for as long as the journal or repository allows.
Access Criteria: Access request will include a description of the research that justifies the use of resources, a research objective and design that described the hypothesis and approach, an analysis plan that includes security safeguards to the data, and a research use statement to be made publicly available. Requesting investigators must sign a Data use Agreement for research data and requestors must have IRB clearance or exemption from their institution. University of Hawaii at Manoa (UHM) Single Entity IRB approval will provide a clear statement identifying all restrictions or limitations on the use of distribution of research materials. The research data submitted to NIH will have proper documentation to ensure meaningful use of data. The study documentation will be in electronic format, comprehensive, and clear to enable investigators to understand the study and data.